CLINICAL TRIAL: NCT04562298
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LCAR-M23, a CAR-T Cell Therapy Targeting MSLN in Patients With Relapsed and Refractory Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study.
Sponsor: Shanghai East Hospital (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry); East Clinical Center of Oncology (Unknown); Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L201906
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-10

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-M23 Chimeric Antigen Receptor T cell (Experimental)
  Interventions: Biological: LCAR-M23 cells

INTERVENTIONS:
Biological: LCAR-M23 cells — Prior to infusion of LCAR-M23, subjects will receive a premedication regimen (intravenous infusion of cyclophosphamide 300 mg/m2 and fludarabine 30 mg/m2 once daily for 3 days; fludarabine dose reduction to 25 mg/m2 and cyclophosphamide to 250 mg/m2 are allowed if the subject' s creatinine clearance is 50-70 mL/min/1.73 m2). A single dose, single Infusion of LCAR-M23 is scheduled 5 to 7 days after the initiation of the premedication regimen.

SUMMARY:
This study is a prospective, single-arm, open-label, single-dose dose finding and extension study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy profiles of the LCAR-M23 CAR-T cell therapy in subjects with relapsed and refractory epithelial ovarian cancer after prior adequate standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects have been fully informed of the possible risks and benefits of participating in this study and have voluntarily signed the informed consent form (ICF)
2. Age: 18-70 years (including 18 and 70 years)
3. Female subjects with histologically or cytologically confirmed advanced epithelial ovarian cancer including fallopian tube and primary peritoneal cancers
4. Mesothelin (MSLN) positive
5. Prior adequate standard of care, treatment failure or intolerance.
6. Imaging shows an evaluable tumor lesion
7. ECOG 0-1
8. Expected survival ≥ 3 months

Exclusion Criteria:

1. Patients who have received the following anti-tumor treatments prior to apheresis:

   * Cytotoxic therapy within 14 days
   * Small molecule targeted therapy within 14 days or at least 5 half-lives, whichever is shorter
   * Therapy with monoclonal antibody within 21 days
   * Immunomodulatory therapy within 7 days
   * Radiotherapy within 14 days and endocrine therapy within 14 days (including tamoxifen, aromatase inhibitor, high-potency progesterone and gonadotropin-releasing hormone analogue, etc.)
2. Previously treated with CAR-T/TCR-T cell therapy against any target or other cell therapies or therapeutic tumor vaccine
3. Previously treated with any MSLN-targeted therapy
4. Brain metastases with central nervous system symptoms
5. Pregnant or lactating women
6. Any condition in which, in the opinion of the investigator, the subject is ineligible for participation in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and incidence, severity, and type of treatment-emergent adverse events (TEAEs) | 90 days post infusion
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose. An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
MTD/ RP2D regimen finding | 90 days post infusion
  Maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D)
Chimeric Antigen Receptor T (CAR-T) Positive Cell Concentration | 2 years post infusion
  Venous blood samples will be collected for measurement of CAR-T positive cellular concentration

SECONDARY OUTCOMES:
Disease control rate (DCR) after administration | 2 years post infusion
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response, partial response and stable disease.
Objective Response Rate (ORR) after administration | 2 years post infusion
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LCAR-M23 cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease as per RECIST 1.1 criteria only.
Time to Response (TTR) after administration | 2 years post infusion
  Time to Response (TTR) is defined as the time interval from the date of first infusion of LCAR-M23 cell formulation to the date of the first response evaluation of the subject who has met all criteria for PR or better.
Duration of Response (DOR) after administration | 2 years post infusion
  Duration of Response (DOR) is defined as the time from the first documentation of response (PR or better) to the first documentation of disease progression evidence (as per RECIST 1.1 criteria) of the responders (who achieve PR or better response).
Progress Free Survival (PFS) after administration | 2 years post infusion
  Progression Free Survival (PFS) is defined as the time interval from the date of first infusion of LCAR-M23 cell formulation to the first documentation of disease progression (as per RECIST 1.1 criteria) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | 2 years post infusion
  Overall survival (OS) is defined as the time interval from the date of first infusion of LCAR-M23 cell formulation to death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, PhD, Principal Investigator — East Clinical Center of Oncology; Yu Kang, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China